CLINICAL TRIAL: NCT02368106
Title: Patient Registry for Prospective Research on Evolving Radiation Oncology Techniques and Quality
Brief Title: Prospective Patient Registry for Radiation Oncology Techniques and Quality
Acronym: GCC 1490
Status: Withdrawn | Type: Observational
Why Stopped: PI decision
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principle Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00060494
Record Dates: First submitted 2015-01-20; First posted 2015-02-20 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumors; Cancer
Keywords: patient registry; radiation oncology; technology assessment
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiation Therapy: Participants receiving one of the 11 listed therapy modalities.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — targeted radiation treatment

SUMMARY:
This study will create a patient data registry to collect and analyze information on technology usage and outcomes among patients receiving a broad range of relatively new radiation treatments that have become standards of care in our practice. Review of this information will serve as a basis for development of better patient management plans, to inform decisions about acquisition of new technologies, to provide information about quality in our care delivery, and to create a database that will securely warehouse ongoing information about what treatments the patients we serve need most and the challenges they face in the treatment process. The information gathered is likely to not only improve our services at the University of Maryland and its community sites but to advance medical science and enhance the quality of care for cancer patients.

DETAILED DESCRIPTION:
The purpose of this study is to create a robust and long-term patient data registry containing limited demographic, diagnostic, treatment, and follow-up data on patients at the study sites undergoing one or more of the following radiation treatments/technologies:

Brachytherapy, including High-Dose-Rate and Low-Dose-Rate Techniques/ GammaPod Therapy/ GRID Treatment/ Image-Guided Radiation Therapy/ Intensity-Modulated Radiation Therapy and Intensity-Modulated Arc Therapy/ MammoSite and SAVI Applicator/ Photodynamic Therapy/ Proton Therapy/ SIR Spheres and Radiolabeled Microsphere Therapy/ Stereotactic Radiosurgery and Stereotactic Body Radiotherapy/ Thermal Therapy (Hyperthermia)

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years old or older and scheduled to undergo any of the listed radiation treatment technologies at the University of Maryland Medical Center or one of its community sites as included in this protocol provided s/he consents to participate.

Exclusion Criteria:

* Patients who are incarcerated or in legal custody are not eligible for this study.
* Patients who are younger than 18 years, are cognitively impaired, or are otherwise unable to provide informed consent.
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Numbers of patients experiencing toxicities/adverse events both during and at follow-up after radiation therapy with any of 11 therapeutic modalities. | 5 years
  Records will be assessed to identify per-patient numbers and grades of toxicities and adverse events resulting from radiation treatment for oncologic conditions as graded by treating physicians according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) during the period of radiation treatment and at each regularly scheduled clinical follow-up appointment, for each of the 11 therapeutic modalities listed as interventions.

SECONDARY OUTCOMES:
Numbers of patients with different initial diagnoses associated with short- and long-term toxicities with specific radiation treatments. | 5 years
  Records will be assessed to identify numbers of patients with specific initial diagnoses (from approximately 100 International Statistical Classification of Diseases and Related Health Problems [ICD 9] malignant neoplasm diagnoses) who experience short- and long-term toxicities after any of the 11 therapeutic modalities listed as interventions.
Numbers of men and women who experience short- and long-term toxicities after specific radiation treatments. | 5 years
  Records will be assessed to identify numbers of men and women who experience CTCAE-defined levels of toxicity during and after radiation treatment with any of the 11 therapeutic modalities listed as interventions.
Age differences in short- and long-term toxicities associated with specific radiation treatment modalities. | 5 years
  Records will be assessed to identify numbers of men and women between the ages of 18-30, 31-40, 41-50, 51-60, 61-70, 71-80, 81-90, and ≥90 years who experience CTCAE-defined levels of toxicity during and after radiation treatment with any of the 11 therapeutic modalities listed as interventions.
Patient income differences in short- and long-term toxicities associated with specific radiation treatment modalities. | 5 years
  Records will be assessed for income (by patient home zip code per U.S. Internal Revenue statistics available at http://www.irs.gov/uac/SOI-Tax-Stats-Individual-Income-Tax-Statistics-ZIP-Code-Data-(SOI)) to identify income level differences and per-patient numbers/ types of CTCAE-defined levels of toxicity during and after radiation treatment with any of the 11 therapeutic modalities listed as interventions.

CONTACTS AND LOCATIONS:
Overall Officials: William Regine, MD, Principal Investigator — UMMC MSGCC Department of Radiation Oncology
Locations (1):
- Ummc Msgcc, Baltimore, Maryland, United States